CLINICAL TRIAL: NCT04161781
Title: Pilot Trial of 18F-BMS-986229 PET in Esophagogastric Cancer
Brief Title: A Study of PET Scans With the Radioactive Tracer 18F-BMS-986229 in Patients With Esophageal, Stomach, or Gastroesophageal Junction Cancer
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: 19-122
Record Dates: First submitted 2019-11-12; First posted 2019-11-13 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2024-03

CONDITIONS: Esophagogastric Cancer; Esophagus Cancer; Esophageal Cancer; Gastric Cancer; Gastric Adenocarcinoma; Gastroesophageal Junction Adenocarcinoma; Gastroesophageal Junction Squamous Cell Carcinoma
Keywords: 18F-BMS-986229; Memorial Sloan Kettering Cancer Center; 19-122
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms | interventions — Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- Cohort 1: 10 participants will receive one injection of 18F-BMS-986229 (370 MBq) and will then undergo whole-body PET/CT (80 mA) encompassing the vertex of the skull to the proximal thigh performed at 60 minutes (within the range of 55-70 minutes) postinjection. The scan itself is expected to last about 30 minutes and participants will be asked to remain in the waiting area or dedicated room for an additional 30 minutes post scan. The total time from injection will be 120 minutes. In both cohorts, participants whose treatment includes nivolumab and who have positive tumor localization observed at baseline will be asked to undergo an additional round of imaging.
  Interventions: Drug: 18F-BMS-986229 Injection; Diagnostic Test: PET/CT Scan
- Cohort 2: 25 participants may receive 370 MBq of 18F-BMS-986229 given intravenously and will undergo a single PET/CT scan 60 minutes (within the range of 55-70 minutes) postinjection. The scan itself is expected to last about 30 minutes and participants will be asked to remain in the waiting area or dedicated room for an additional 30 minutes post scan. The total time from injection will be 120 minutes. In both cohorts, participants whose treatment includes nivolumab and who have positive tumor localization observed at baseline will be asked to undergo an additional round of imaging. If the participant agrees, they will receive a second injection while undergoing nivolumab treatment (after at least 2 cycles or 6 weeksof therapy).
  Interventions: Drug: IV 18F-BMS-986229; Diagnostic Test: PET/CT Scan

INTERVENTIONS:
Drug: 18F-BMS-986229 Injection — Single injection prior to scan
  Groups: Cohort 1
Drug: IV 18F-BMS-986229 — 370 MBq administered intravenously prior to scan
  Groups: Cohort 2
Diagnostic Test: PET/CT Scan — Whole-body PET/CT (80 mA)

SUMMARY:
The purpose of the study is to test 18F-BMS-986229 positron emission tomography (PET) imaging a practical and safe way to check the status of esophageal, stomach, and gastroesophageal junction cancer.

ELIGIBILITY:
Inclusion Criteria:

* Participant must have pathologically or cytolofically confirmed (at MSK) esophageal, gastric, or gastroesophageal junction adenocarcinoma or squamous cell carcinoma
* PD-L1-positive expression in >/=1% of the tumor or stromal cells. PD-L1 expression will be reviewed by MSK pathologist, scored and recorded using the combined positive score (CPS) formula (number of PD-L1 positive tumor cells, lymphocytes, and macrophages divided by the number of tumor cells x 100).
* Participants must have disease that can be evaluated radiographically. This may be measurable disease or nonmeasurable disease according to RECIST 1.1.
* Concurrent therapy is allowed.
* Age 18 years or older.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
* Female subjects of childbearing potential must have a negative urine or serum pregnancy test within 24 hours before receiving the first dose of the study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Adequate organ function, as defined in Table 1. All screening labs should be performed within 14 days of initiation of treatment.

Hematological Absolute neutrophil count: >/=1,000/mCL Platelets: >/=90,000/mCL Hemoglobin: >/=8 g/dL

Renal Serum creatinine: </=2.0 x upper limit of normal (ULN)

Hepatic Serum total bilirubin: </=2.5 x ULN (1.5 mg/dL or 25.65 umol/L) OR (except patients with Gilbert's disease [</=3 x ULN]) AST (SGOT) and ALT (SGPT): </=2.5 x ULN OR </=5 x ULN for subjects with liver metastases

Exclusion Criteria:

* Known diagnosis of immunodeficiency or receipt of systemic steroid therapy or any other form of immunosuppressive therapy within 7 days before the first dose of trial treatment
* History of active tuberculosis (Bacillus tuberculosis)
* Active or documented autoimmune or inflammatory disorder (including inflammatory bowel disease, systemic lupus erythematous, Wegener syndrome [granulomatosis with polyangitis], myasthenia gravis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis) within the 3 years before the start of treatment. The following are exceptions to this criterion:

  * Subjects with vitiligo or alopecia
  * Subjects with hypothyroidism (e.g., following Hashimoto syndrome) who are stable with hormone replacement therapy or with psoriasis not requiring systemic treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potential research subjects will be identified by members of the patient's treatment team, the protocol investigator or research team. If the investigator is a member of the treatment team, s/he will screen their patient's medical records for suitable research study participants. The investigator will use information provided by the patient and/or medical record to confirm that the patient is eligible and contact the patient regarding study enrollment. All eligible patients, regardless of sex and race will be approached for participation. No additional measures, e.g. advertisement, payment to patients, will be employed to recruit patients.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2019-11-12 (Actual); Primary Completion 2024-03-06 (Actual); Study Completion 2024-03-06 (Actual)

PRIMARY OUTCOMES:
Feasibility of 18F-BMS-986229 PET in participants with Gastroesophageal Cancer | 4 weeks
  18F-BMS-986229 PET will be considered feasible if there are no Grade 3 or higher 18F-BMS-986229 related adverse events and if at least 7 to 10 participants in Cohort 1 (70%) are found to be 18F-BMS-986229 PET positive.

CONTACTS AND LOCATIONS:
Overall Officials: Yelena Janjigian, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- [Derived] Cytryn SL, Pandit-Taskar N, Lumish MA, Maron SB, Gu P, Ku GY, Chou JF, Capanu M, Antoine A, Loegel D, Feder L, Philemond S, Lyashchenko SK, Lewis JS, Paroder V, Srivastava A, Tang LH, Schoder H, Janjigian YY. 18F-BMS-986229 PET to Assess Programmed-Death Ligand 1 Status in Gastroesophageal Cancer. J Nucl Med. 2024 May 1;65(5):722-727. doi: 10.2967/jnumed.123.267186. PMID 38514081
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org